CLINICAL TRIAL: NCT07144514
Title: A Retrospective Observational Study Investigating Demographic and Clinical Characteristics of SLE Patients in Egypt: Unveiling the Burden, Reasons for Hospitalization, and ER Visits in Participating Centers
Brief Title: Observational Study Investigating Demographic and Clinical Characteristics of SLE Patients in Egypt
Acronym: ROSE
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00088
Record Dates: First submitted 2025-05-13; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systemic lupus erythematosus (SLE) is an autoimmune condition characterized by a complicated, unclear etiology that involves various complex factors. SLE symptoms and indications are broadly classified as organ-specific and constitutional (arising from systemic inflammation). While fever, weight loss, and elevated body temperature are constitutional symptoms that patients with SLE may encounter, SLE may affect specific organs, including the lungs, heart, kidneys, and muscles, as well as the hematologic and central nervous systems. If left untreated, SLE-related local inflammation may result in permanent organ damage. Individuals diagnosed with SLE frequently encounter instances of heightened disease activity, commonly referred to as disease exacerbations or flares. Flares are described as "a distinct surge in disease activity affecting one or more organ systems, as demonstrated by an onset of novel or worsening clinical symptoms and/or laboratory findings". Due to the complex trajectory of SLE, patients may have a higher likelihood of visiting the emergency room (ER) because of flare-ups, adverse drug reactions, and noncompliance with prescribed treatment regimens. Furthermore, SLE has a high cumulative morbidity and mortality rate, and comorbidities linked to the disease have become a major cause of late deaths in SLE. Although the prevalence of SLE varies by age, gender, and geographical distribution, the global prevalence of SLE was estimated to be 43.7% (15.87 to 108.92) per 100,000 individuals and 3.41 million individuals for the entire population. A recent study by Gheita et al. estimated the prevalence of SLE among adults in Egypt to be 6.1 per 100,000; however, the researchers highlighted the scarcity of published epidemiological studies on the Egyptian SLE patient population, and the available data is based mostly on single-center studies with small sample sizes. Thus, the available data is not representative of the whole nation. This study aims to overcome these issues and address the data gap regarding the SLE patient population in Egypt.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of both genders aged 18 or older at the time of study inclusion.
2. Patients with medical records from the selected sites between 2016 and 2023 with at least one year of follow-up records.
3. Patients receiving routine treatment in the participating sites.
4. Patients with an SLE diagnosis.
5. Due to the retrospective nature of the study a waiver grant of the consent will be requested from the IRB/IEC for the study participants, if waiver not granted Patient or next of kin/legal representative (for deceased patients at study entry) willing and able to provide written informed consent according to the local regulations.

Exclusion Criteria:

1. Patients with new-onset SLE as they will have insufficient data.
2. Patients whose records have insufficient data (for example, due to lost follow up).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include adult patients diagnosed with SLE in different geographic areas of Egypt who meet all the specified inclusion criteria and none of the exclusion criteria for this study. The study population should be selected without bias.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Description of the lupus-affected population | 60 months
  patients gender, age, and percentage of patients with affected organs, as well as medications taken.
Determining the burden of SLE in Egypt | 60 months
  The average number of SLE flares

SECONDARY OUTCOMES:
Mortality rate | 60 Months
  Percentage of mortality within the duration of data collection and reason for mortality (all-cause mortality, SLE-related manifestation, mortality due to comorbidities or medications).

OTHER OUTCOMES:
Description of treatment lines | 60 Months
  The duration of each treatment line and any observed outcomes
Determining the disease progression of SLE involves assessing and understanding how the condition evolves and changes over time | 60 Months
  The proportion and percentage of patients suffering from an increase/emergence of SLE manifestations